CLINICAL TRIAL: NCT04894292
Title: Adverse Obstetrical Outcomes for Women With Adenomyosis
Brief Title: The Effect of Adenomoyosis on Pregnancy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ahkam Göksel Kanmaz, Assoc. Prof, Tepecik Training and Research Hospital
Other Study IDs: TepecikTRH-001
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Adenomyosis; Pregnancy Complications
Keywords: adenomyosis; pregnancy complications; MUSA classification; ultrasound
MeSH Terms: conditions — Adenomyosis; Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adenomyosis Group
  Interventions: Other: Non intervention
- Non-adenomyosis Group
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — During the study there is no extra intervention planned for the participants.

SUMMARY:
Adenomyosis can be defined as the settling of endometrial gland cells in the myometrium and deformity in the uterus and the prevalence of adenomyosis is according to the patient population and countries around 20%. There are recent publications reporting that this rate increases up to 50% in women dealing with infertility. In adenomyosis, where uterine morphology is affected, it is not thought that the uterus, which is expected to provide many morphological adaptations during pregnancy, will not be affected. Therefore, in this prospective study, it was planned to investigate the effects of adenomyosis during pregnancy.

For this study the presence of adenomyosis will be questioned by using ultrasonographic morphological uterine limitation (MUSA) in women who apply to the outpatient clinic with suspicion of pregnancy and undergo transvaginal ultrasonography for the diagnosis of pregnancy before sixth gestational week.

Patients will be divided into two groups according to the presence of adenomyosis and pregnancy complications such as preterm labor, premature rupture of membranes, cesarean section rates, preeclampsia, fetal malpresentation and preeclampsia will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 years
* Being diagnosed before the 6th gestational week
* Having all pregnancy follow-ups and deliveries in our hospital

Exclusion Criteria:

* Previous uterine surgery
* Multiple pregnancies
* Pregnant women with uterine malformations
* Pregnant women with fetal anomalies
* Those who got pregnant using assisted reproductive technique

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women diagnosed by TV usg before the 6th gestational week will be divided into two according to the MUSA classification, and those with adenomyosis who are not in the study group will be evaluated as the control group.
  All the participants should be at between 18-35 age years old and all perinatal visits and deliveries should be at Tepecik Obstetric Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy complication | 15 month
  Preterm labour

SECONDARY OUTCOMES:
Pregnancy complication | 16 month
  placental anomalies
Pregnancy complication | 17 month
  preeclampsia, eclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Ahkam Göksel Kanmaz, Assoc. Prof., Study Director — Tepecik Education and Research Hospital
Locations (1):
- Tepecik Education and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harada T, Taniguchi F, Amano H, Kurozawa Y, Ideno Y, Hayashi K, Harada T; Japan Environment and Children's Study Group. Adverse obstetrical outcomes for women with endometriosis and adenomyosis: A large cohort of the Japan Environment and Children's Study. PLoS One. 2019 Aug 2;14(8):e0220256. doi: 10.1371/journal.pone.0220256. eCollection 2019. PMID 31374085
- [Background] Horton J, Sterrenburg M, Lane S, Maheshwari A, Li TC, Cheong Y. Reproductive, obstetric, and perinatal outcomes of women with adenomyosis and endometriosis: a systematic review and meta-analysis. Hum Reprod Update. 2019 Sep 11;25(5):592-632. doi: 10.1093/humupd/dmz012. PMID 31318420